CLINICAL TRIAL: NCT05068843
Title: Arthroscopic Partial Meniscectomy Versus Physical Therapy for Patients Over 45 Years With a Meniscal Tears: 5-year Follow-up of the ESCAPE Trial
Brief Title: Arthroscopic Partial Meniscectomy Versus Exercise Therapy for Meniscal Injuries in Older Patients, a 5 Year Follow up.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Responsible Party: Principal Investigator, Rudolf W Poolman, MD PhD, Principal Investigator, Onze Lieve Vrouwe Gasthuis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2021-02-23; First posted 2021-10-06 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Meniscus Tear, Tibial; Osteoarthritis, Knee
MeSH Terms: conditions — Tibial Meniscus Injuries; Osteoarthritis, Knee | interventions — Physical Therapy Modalities; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthroscopic partial meniscectomy (Active Comparator): In the surgery group, the orthopaedic surgeon performed an arthroscopic partial meniscectomy (APM) within 4 weeks after allocation. The surgeon removed the damaged part of the meniscus, until a stable and solid meniscus remained. All patients received written post-operative instructions. Eight weeks after surgery, patients received a consult in the outpatient orthopaedic clinic. In agreement with the Dutch Orthopaedic Association Guidelines, patients were referred to physical therapy when signs of abnormal recovery were present.
  Other Names:
  APM meniscal surgery surgery
  Interventions: Procedure: arthroscopic partial meniscectomy
- Physical therapy (Other): The physical therapy program consisted of a physical therapist-led incremental exercise program containing of coordination/balance, closed kinetic chain strengths and cardiovascular exercises (see Appendix 1). The program was designed for 8 weeks with a total of 16 treatment sessions, each with a duration of 30 minutes. All 16 sessions were reimbursed. If knee symptoms persisted following the physical therapy program (e.g., knee pain, limitations in daily activities or mechanical dysfunction ), the patient could attend additional physical therapy sessions (not reimbursed by the study) or have meniscal surgery, depending on a shared decision after consultation with their orthopaedic surgeon.
  Interventions: Other: Physical therapy

INTERVENTIONS:
Procedure: arthroscopic partial meniscectomy — In the surgery group, the orthopaedic surgeon performed an arthroscopic partial meniscectomy within 4 weeks after allocation. The surgeon removed the damaged part of the meniscus, until a stable and solid meniscus remained. All patients received written post-operative instructions. Eight weeks after surgery, patients received a consult in the outpatient orthopaedic clinic. In agreement with the Dutch Orthopaedic Association Guidelines, patients were referred to physical therapy when signs of abnormal recovery were present.
  Other Names: meniscal surgery; APM
  Arms: Arthroscopic partial meniscectomy
Other: Physical therapy — The treatment protocol consisted of a physical therapist-led incremental exercise program over a period of eight weeks, containing 16 sessions of 30 minutes each.
  Other Names: exercise therapy
  Arms: Physical therapy

SUMMARY:
Arthroscopic partial meniscectomie (APM) offers little short-term to medium-term benefit above sham surgery or non-surgical management for knee function in most patients with a symptomatic degenerative meniscus tear. It is suggested that APM is associated with increased risk of accelerated progression of knee osteoarthritis in middle-aged to older patients.

With the 5 year follow-up of the ESCAPE trial we will investigate the longterm results of APM and physical therapy in patients with a meniscal tear over 45 years old.

ELIGIBILITY:
Inclusion Criteria:

* 45 to 70 years old MRI confirmed, non-obstructive and symptomatic meniscal tear

Exclusion Criteria:

* Knee locking or trauma leading to acute surgery;

  ▸ Associated injuries on the index knee consisting of:
* Symptomatic partial or total tear of the anterior cruciate ligament (ACL),
* Posterior cruciate ligament tear,
* OA of the knee, grade 4 on the Kellgren and Lawrence Grading Scale,
* An injury to the lateral or posterolateral ligament complex with significant laxity;

  * Previous knee surgery on the index knee (with the exception of diagnostic arthroscopy);
  * Tumour that is suspected of malignancy, detectable on MRI;
  * Obesity with a body mass index >35;
  * American Society of Anesthesiologists (ASA) class 4 or 5 patients;
  * General disease that effects physical function or systemic medication/abuse of steroids;
  * Any other medical condition or treatment interfering with the completion or assessment of the trial, for example, contraindications to MRI or surgery;
  * Drugs or alcohol abuse;
  * Patients unable to fill out the Dutch questionnaires.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2013-07-13 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Knee Documentation Committee Subjective Knee Form (IKDC) questionnaire | 60 months
  Knee Documentation Committee Subjective Knee Form (IKDC) questionnaire to assess patient reported knee functionWe assessed knee OA on radiographs and patient reported frequency of knee pain during activities was assessed as part of the IKDC questionnaire.

SECONDARY OUTCOMES:
Radiographic Knee osteoarthritis | 60 months
  The OARSI atlas is a semi-quantitative instrument with focus to assess the severity of joint space narrowing and osteophytes in knee OA. We considered radiographic knee OA if any of the follow three criteria were met: 1) Joint space narrowing of grade 2 or higher; 2) sum of osteophyte grades ≥2 or 3) grade 1 joint space narrowing in combination with a grade 1 osteophyte.
Symptomatic knee osteoarthritis (OA) | 60 months
  Our main outcome is symptomatic knee osteoarthritis (OA). Symptomatic knee OA is a combination of knee OA assessed on radiograph and patient reported frequency of knee pain.
  We assessed knee OA on radiographs and patient reported frequency of knee pain during activities was assessed as part of the IKDC questionnaire.
Patient reported knee pain during weight bearing | 60 months
  Patient reported knee pain during weight bearing assessed on visual analogue scale from 0-100
Patient reported quality of life | 60 months
  Quality of life assessed by the Euroqol 5 diminesions 5 Levels

IPD SHARING:
Plan to Share IPD: Yes
available on request